CLINICAL TRIAL: NCT00962585
Title: Randomized, Double Blind, Multicenter, Placebo Controlled, Proof of Concept Trial to Assess the Efficacy and Safety of 4 Weeks Treatment With AUS-131 (S-equol) on Vasomotor Symptoms in Menopausal Patients
Brief Title: Efficacy and Safety of S-equol on Vasomotor Symptoms in Menopausal Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ausio Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AUS-CT03
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Results first posted 2014-04-08 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-03

CONDITIONS: Menopause
MeSH Terms: interventions — Equol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- S-equol 10 mg BID (Experimental): S-equol 20 mg total daily dose
  Interventions: Drug: S-equol
- S-equol 50 mg BID (Experimental): S-equol 100 mg total daily dose
  Interventions: Drug: S-equol
- S-equol 150 mg BID (Experimental): S-equol 300 mg total daily dose
  Interventions: Drug: S-equol

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: S-equol — Eligible patients meeting all study entry criteria were randomly assigned to receive one of the following active treatments for 4 weeks:
  * S-equol 10 mg BID (20 mg total daily dose)
  * S-equol 50 mg BID (100 mg total daily dose)
  * S-equol 150 mg BID (300 mg total daily dose)
  Other Names: AUS-131
  Arms: S-equol 10 mg BID; S-equol 150 mg BID; S-equol 50 mg BID

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of S-equol in menopausal patients with hot flushes and night sweats.

DETAILED DESCRIPTION:
The study is a randomized, double blind, multicenter, placebo controlled, parallel group, proof of concept study comparing the efficacy, safety, and acceptability of 3 doses of S-equol to placebo in menopausal patients with vasomotor symptoms. The study objective is an evaluation of the dose response of 3 dose levels of AUS-131 (S-equol) and placebo with respect to reducing the mean number of moderate to severe vasomotor symptoms after 4 weeks of treatment. The safety of S-equol will be evaluated during the study.

ELIGIBILITY:
Inclusion Criteria:

* 12 months of spontaneous amenorrhea, or 6 months of spontaneous amenorrhea with serum follicle stimulating hormone (FSH) concentrations > 40 mIU/mL, or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy, or hysterectomy with 2 (measured 14 days apart) serum FSH concentrations > 40 mIU/mL.
* Is likely to experience at least 50 moderate to severe vasomotor symptoms ([MSVS] hot flushes and nocturnal sweating) per week while not receiving estrogen replacement therapy based on history of menopause, in the judgment of the investigator.
* Documented experiencing at least 50 MSVS per week during the 14 day baseline period before the Randomization Visit (Visit 3), based on the patient diary entries (calculated mean MSVS/week for the 14 day baseline period).
* If ≥ 40 years of age, has a documented negative mammogram and a normal clinical breast examination with no findings indicative of breast malignancy.
* Has a body mass index (BMI) < 35.0 kg/m2.

Exclusion Criteria:

* Has a known history of allergic reaction or clinically significant intolerance to ingredients of the study drug.
* Received any of the following:oral or dermal estrogen/progestin or selective estrogen receptor modulator (SERM) containing drug product therapy within 8 weeks before Screening, injectable or implantable estrogen/progestin therapy within 3 months before Screening, hormone releasing intrauterine device
* Had unexplained or otherwise abnormal vaginal bleeding within 6 months before Screening.
* Has a history of, or currently has, any of the following conditions: thrombophlebitis, thromboembolic disease, estrogen dependent neoplasia, or carcinoma of the breast.
* Has a history of any untreated or uncontrolled endocrine disorders (e.g., hyperparathyroidism, uncontrolled hyperthyroidism).
* Has any clinically significant unstable cardiac, respiratory, neurological, immunological, hematological, hepatic, renal, endocrine, or gastric disease or any other condition that, in the opinion of the investigator, could compromise the patient's welfare, ability to communicate with the study staff, or otherwise contraindicate study participation.
* Has clinically significant depression or severe psychiatric disturbances.
* Has active liver disease with aspartate aminotransferase (AST) > 3 times the upper limit of normal (ULN), alanine aminotransferase (ALT) > 3 times ULN, unexplained alkaline phosphatase > 3 times ULN, total bilirubin > 2 times ULN, renal insufficiency with creatinine > 1.7 mg/dL, or clinically significant abnormal hemoglobin, white blood cell count, or platelet count.
* Has an endometrial thickness ≥ 4 mm.
* Has a history indicative of endometrial hyperplasia or cancer.
* Shows presence of any manifest premalignant or malignant disease except treated skin cancers (except melanoma).
* Has known or suspected history of alcoholism or drug abuse or misuse within the past 5 years.
* Has resting systolic blood pressure (BP) > 160 mmHg or < 90 mmHg, or diastolic BP > 90 mmHg or < 60 mmHg at Screening.
* Has a history of smoking more than 5 cigarettes daily within the year before Screening.
* Has tested positive on the urine drug screen. Patients who test positive at Screening and can produce documentation from their physician for the medication that caused the positive test may be considered for study enrollment at the discretion of the investigator.
* Has significant difficulties swallowing capsules or is unable to tolerate oral medication.
* Has participated in another clinical trial or received any investigational drug or device or investigational therapy within 30 days before Screening.
* Has a disorder that affects gastrointestinal absorption.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Thomas, MD, Principal Investigator — University of Cincinnati
Locations (9):
- United States (5):
  - Bluegrass Clinical Research, Louisville, Kentucky
  - Greater Cincinnati OB/GYN, Inc., Cincinnati, Ohio
  - Rapid Medical Research, Cleveland, Ohio
  - Radiant Research, Inc, Greenville, South Carolina
  - Advanced Clinical Research, West Jordon, Utah
- Australia (4):
  - Sydney Centre for Reproductive Health Research, Ashfield, New South Wales
  - Royal Hospital for Women, Randwick, New South Wales
  - Women's Health Center, Royal Adelaide Hospital, Adelaide, South Australia
  - Emeritus Research, Malvern East, Victoria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients for this trial were screened from 9 investigative sites in the United States and Australia. Participants were women of menopausal status and experiencing vasomotor symptoms and nocturnal sweating.
Pre-assignment Details: After completing screening visit assessments, subjects were instructed to refrain from taking prohibited medications throughout the study. Patients who were taking prohibited medications at the time of the screening visit discontinued their use and completed a suitable washout period before progressing to the next visit.
Groups:
- S-equol 10 mg BID: 20 mg total daily dose of S-equol
- S-equol 50 mg BID: 100 mg total daily dose of S-equol
- S-equol 150 mg BID: 300 mg total daily dose of S-equol
- Placebo: Placebo treatment arm
Period: Overall Study
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo
Started | 43 | 42 | 42 | 42
Completed | 37 | 40 | 39 | 42
Not Completed | 6 | 2 | 3 | 0
Not completed — Adverse Event | 0 | 2 | 1 | 0
Not completed — Lost to Follow-up | 3 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Withdrew Consent | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo | Total
Number analyzed (Participants) | 43 | 42 | 42 | 42 | 169
Age, Customized [Mean (Standard Deviation); unit: years] | 53.8 (7.9) | 53.1 (6.9) | 54.9 (5.8) | 56.2 (6.7) | 54.5 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 42 | 42 | 42 | 169
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 0 | 0 | 1 | 1
  Black or African American | 4 | 7 | 10 | 5 | 26
  White | 39 | 35 | 32 | 34 | 140
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2
Height [Mean (Standard Deviation); unit: centimeters] | 165.3 (5.1) | 164.1 (4.6) | 165.4 (6.7) | 163.3 (5.9) | 164.5 (5.6)
Weight [Mean (Standard Deviation); unit: kilograms] | 74.1 (11.6) | 73.0 (10.7) | 74.4 (10.1) | 73.2 (12.8) | 73.7 (11.3)
Body Mass Index [Mean (Standard Deviation); unit: kilogram/meter^2] | 27.1 (3.9) | 27.1 (4.1) | 27.2 (3.5) | 27.4 (4.1) | 27.2 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Frequency of Moderate to Severe Vasomotor Symptoms (MSVS) Baseline at Week 4 (2-week Period)
Description: The primary efficacy endpoint for this study was the change from Baseline (Day 0) in the frequency of MSVS (difference between Baseline [2-week run-in period] and Week 4), where the baseline MSVS frequency was captured over 14 ± 2 day period. Moderate is defined as "sensation of heat with sweating, able to continue activity"; severe is defined as "sensation of heat with sweating, causing cessation of activity". Patients used the take-home daily diary to record MSVS information during the run-in period and treatment period and analyses were performed as specified.
  Treatment group differences are estimated using least squares (LS) means and 95% confidence intervals based on the mean square error from the ANCOVA. LSMeans refer to overall adjusted mean frequency of MSVS.
Time Frame: 4 weeks from Baseline (2-week run-in period)
Population: The analysis population consists of all randomized patients who received at least 1 dose of randomized study drug starting at visit 3, who had at least 1 post-dose efficacy assessment. Missing efficacy data were not imputed.
Measure: Mean (95% Confidence Interval); unit: Number of MSVS/2 weeks
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo
Number analyzed (Participants) | 42 | 42 | 41 | 42
Number of MSVS/2 weeks
  Baseline (Day 0) | 73.5 [65.3 to 81.8] | 69.5 [64.0 to 75.1] | 70.4 [63.5 to 77.3] | 67.9 [61.4 to 74.4]
  Week 4 | 41.7 (32.8) [31.0 to 52.5] | 46.1 (27.8) [37.5 to 54.8] | 39.3 (27.3) [30.5 to 48.0] | 39.3 (25.1) [31.5 to 47.1]
  Change from Baseline at Week 4 | -30.1 (29.0) [-39.7 to -20.6] | -23.4 (30.2) [-32.8 to -14.0] | -31.1 (23.4) [-38.6 to -23.7] | -28.6 (22.1) [-35.5 to -21.7]
  LSMean | 40.78 [32.72 to 48.84] | 46.63 [38.87 to 54.39] | 40.59 [32.58 to 48.59] | 39.65 [31.89 to 47.41]
Statistical Analysis 1: Comparison: S-equol 10 mg BID vs S-equol 50 mg BID vs S-equol 150 mg BID vs Placebo; # of MSVS per week at each protocol visits = (# of Moderate+Severe hot flushes)/(Current protocol visit date-Previous protocol visit date (days)) x 7. The ANCOVA procedure was used to test the following hypotheses: H0: μ1 = μp versus HA: μ1 ≠ μp where μ1 and μp denote the mean frequency of MSVS (at Week 4 in case of primary efficacy endpoint), adjusted for Baseline MSVS values, in the treatment and placebo groups, respectively; Test type: Superiority or Other; p = 0.5730, ANCOVA — P-value was not adjusted for multiple comparisons and the a priori threshold for statistical significance was P <0.05; Model (Analysis of covariance): Week 4 = Baseline (MSVS) + Treatment + Site Difference Between Means: S-equol treatment group - Placebo
Statistical Analysis 2: Comparison: S-equol 10 mg BID vs Placebo; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = 1.13, 95% CI 2-sided [-10.06 to 12.32]
Statistical Analysis 3: Comparison: S-equol 50 mg BID vs Placebo; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = 6.98, 95% CI 2-sided [-3.87 to 17.84]
Statistical Analysis 4: Comparison: S-equol 150 mg BID vs Placebo; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = 0.94, 95% CI 2-sided [-10.16 to 12.04]

2. Secondary Outcome: Mean Change in Frequency of MSVS From Baseline at Week 4 (1-week Period)
Description: Change from Baseline in the frequency of MSVS (difference between Baseline [period following first 7 days of 2-week run-in period] and period following first 7 days of 2-week Week 4 period), where the Baseline MSVS frequency was captured at visit 3 (Day 0), in the period following the first 7 days, as per CRF. Note: this endpoint is identical to the primary endpoint, however, instead of a 14 ± 2 day period, the period following the first 7 days was used, at Baseline and visit 3.
  Treatment group differences are estimated using least squares (LS) means and 95% confidence intervals based on the mean square error from the ANCOVA. LSMeans refer to overall adjusted mean frequency of MSVS.
Time Frame: 4 weeks from Baseline (period following first 7 days of 2-week run-in period)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Number of MSVS/week
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo
Number analyzed (Participants) | 42 | 42 | 41 | 42
Number of MSVS/week
  Baseline (Day 0) | 73.0 [64.3 to 81.7] | 71.4 [65.4 to 77.4] | 69.5 [62.0 to 76.9] | 67.9 [60.1 to 75.6]
  Week 4 | 40.0 [27.5 to 52.5] | 45.5 [36.3 to 54.6] | 37.1 [28.2 to 46.1] | 40.2 [31.5 to 48.9]
  Change from Baseline at Week 4 | -30.2 [-40.9 to -19.6] | -24.9 [-35.0 to -14.8] | -32.6 [-41.1 to -24.0] | -27.6 [-35.3 to -20.0]
  LSMean | 40.04 [31.02 to 49.06] | 44.99 [36.50 to 53.49] | 38.60 [30.09 to 47.10] | 40.23 [32.00 to 48.45]
Statistical Analysis 1: Comparison: S-equol 10 mg BID vs S-equol 50 mg BID vs S-equol 150 mg BID vs Placebo; # of MSVS per week at each protocol visits = (# of Moderate+Severe hot flushes)/(Current protocol visit date-Previous protocol visit date (days)) x 7 1-week period = remaining days of the period since the last visit (i.e. period following first 7 days, as per CRF); Test type: Superiority or Other; p = 0.7364, ANCOVA — P-value was not adjusted for multiple comparisons and the a priori threshold for statistical significance was P <0.05; Model: Week 4 = Baseline (MSVS) + Treatment + Site Difference Between Means: S-equol treatment group - Placebo
Statistical Analysis 2: Comparison: S-equol 10 mg BID vs Placebo; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = -0.19, 95% CI 2-sided [-12.38 to 12.01]
Statistical Analysis 3: Comparison: S-equol 50 mg BID vs Placebo; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = 4.77, 95% CI 2-sided [-6.94 to 16.48]
Statistical Analysis 4: Comparison: S-equol 150 mg BID vs Placebo; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = -1.63, 95% CI 2-sided [-13.41 to 10.15]

3. Secondary Outcome: Change From Baseline (Day 0) in the Frequency of MSVS at Week 1 and Week 2
Description: The frequency of MSVS per week, at each of the protocol visits, was calculated as follows, for each patient: [# of Moderate+Severe hot flushes)/(Current protocol visit date-Previous protocol visit date (days)] * 7.
  The ANCOVA procedure tested the following hypotheses:
  H0: μ1 = μp versus HA: μ1 ≠ μp, where μ1 and μp denote the mean frequency of MSVS, adjusted for Baseline MSVS values, in the treatment and placebo groups, respectively.
  LSMeans refer to the overall adjusted mean frequecy of MSVS.
Time Frame: 1 and 2 weeks from Baseline (Day 0)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Number of MSVS/week
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo
Number analyzed (Participants) | 42 | 42 | 41 | 42
Number of MSVS/week
  Week 1 | 53.6 [47.4 to 59.8] | 63.1 [55.5 to 70.8] | 54.4 [45.0 to 63.7] | 54.1 [46.6 to 61.6]
  Change from Baseline at Week 1 | -19.9 [-28.6 to -11.2] | -6.7 [-12.7 to -0.7] | -15.9 [-21.6 to -10.2] | -13.8 [-18.8 to -8.8]
  Week 1, LSMean | 50.95 [44.67 to 57.24] | 64.41 [58.04 to 70.78] | 56.03 [49.52 to 62.55] | 54.72 [48.38 to 61.06]
  Week 2 | 47.3 [38.5 to 56.2] | 54.3 [44.2 to 64.4] | 51.0 [40.7 to 61.2] | 50.0 [41.4 to 58.7]
  Change from Baseline at Week 2 | -23.3 [-31.2 to -15.3] | -14.8 [-25.0 to -4.6] | -19.4 [-26.6 to -12.2] | -17.9 [-25.5 to -10.2]
  Week 2, LSMean | 43.96 [35.67 to 52.24] | 54.22 [45.97 to 62.47] | 51.56 [43.21 to 59.92] | 50.66 [42.45 to 58.87]
Statistical Analysis 1: Comparison: S-equol 10 mg BID vs S-equol 50 mg BID vs S-equol 150 mg BID vs Placebo; # of MSVS per week at each protocol visits = (# of Moderate+Severe hot flushes)/(Current protocol visit date-Previous protocol visit date (days)) x 7; Test type: Superiority or Other; p = 0.1217, Repeated measures ANCOVA — P-value was not adjusted for multiple comparisons and the a priori threshold for statistical significance was P <0.05. Treatment effect averaged across Weeks 1 and 2; Mixed Model: MSVS = Baseline (MSVS) + Treatment + Site + Weeks + Treatment x Weeks Difference Between Means: S-equol treatment group - Placebo
Statistical Analysis 2: Comparison: S-equol 10 mg BID vs Placebo; Week 1, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = -3.77, 95% CI [-12.69 to 5.16]
Statistical Analysis 3: Comparison: S-equol 50 mg BID vs Placebo; Week 1, Treatment Effect; Test type: Superiority or Other; p < 0.05, Pair-wise comparisons; LS means difference = 9.69, 95% CI 2-sided [0.79 to 18.60]
Statistical Analysis 4: Comparison: S-equol 150 mg BID vs Placebo; Week 1, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = 1.31, 95% CI 2-sided [-7.73 to 10.36]
Statistical Analysis 5: Comparison: S-equol 10 mg BID vs Placebo; Week 2, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = -6.70, 95% CI 2-sided [-18.36 to 4.96]
Statistical Analysis 6: Comparison: S-equol 50 mg BID vs Placebo; Week 2, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = 3.56, 95% CI 2-sided [-8.01 to 15.14]
Statistical Analysis 7: Comparison: S-equol 150 mg BID vs Placebo; Week 2, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = 0.91, 95% CI 2-sided [-10.77 to 12.58]

4. Secondary Outcome: Change From Baseline (Day 0) in the Severity of VMS as Recorded in the Patient Diary at Week 1, Week 2, and Week 4
Description: The severity of vasomotor symptoms per week at each of the protocol visits was calculated for each patient as follows: [(Sum of scores of Mild, Moderate, Severe hot flushes)/(Current protocol visit date - Previous protocol visit date (days)] * 7, where severity of vasomotor symptoms were scored as: 1 = mild, 2 = moderate and 3 = severe. Higher values represented worse severity.
  LSMeans refer to the overall adjusted mean severity of VMS.
  Hot Flush Classification: Mild: sensation of heat without sweating; Moderate: sensation of heat with sweating, able to continue activity; Severe: sensation of heat with sweating, causing cessation of activity.
  Patients recorded the number of hot flushes (day and night) in their diaries related to the severity (mild/moderate/severe).
Time Frame: 1, 2, and 4 weeks from Baseline (Day 0)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo
Number analyzed (Participants) | 42 | 42 | 41 | 42
units on a scale
  Baseline (Day 0) | 188.6 [168.1 to 209.1] | 177.1 [161.0 to 193.2] | 175.6 [158.8 to 192.4] | 172.8 [155.9 to 189.7]
  Week 1 | 139.0 [123.1 to 155.0] | 160.4 [139.5 to 181.3] | 133.6 [113.9 to 153.4] | 136.0 [116.8 to 155.1]
  Change from Baseline at Week 1 | -49.5 [-66.7 to -32.4] | -17.5 [-32.6 to -2.5] | -41.8 [-55.8 to -27.8] | -36.8 [-48.3 to -25.4]
  Week 1, LSMean | 130.93 [116.79 to 145.07] | 162.94 [148.61 to 177.26] | 139.36 [124.72 to 153.99] | 137.27 [123.02 to 151.52]
  Week 2 | 122.0 [99.5 to 144.5] | 140.1 [114.3 to 165.9] | 126.2 [102.7 to 149.6] | 128.7 [106.3 to 151.1]
  Change from Baseline at Week 2 | -60.4 [-79.2 to -41.7] | -35.3 [-60.4 to -10.2] | -49.4 [-67.3 to -31.6] | -44.1 [-62.1 to -26.2]
  Week 2, LSMean | 113.86 [94.57 to 133.14] | 138.73 [119.57 to 157.89] | 129.34 [109.92 to 148.77] | 130.00 [110.89 to 149.10]
  Week 4 | 110.5 [83.4 to 137.7] | 120.3 [98.0 to 142.6] | 99.5 [78.8 to 120.3] | 101.6 [83.1 to 120.1]
  Change from Baseline at Week 4 | -75.5 [-98.0 to -53.0] | -56.8 [-80.8 to -32.7] | -76.2 [-94.9 to -57.5] | -71.2 [-87.8 to -54.5]
  Week 4, LSMean | 101.27 [81.98 to 120.56] | 119.11 [100.23 to 137.99] | 101.67 [82.39 to 120.94] | 102.96 [84.08 to 121.84]
Statistical Analysis 1: Comparison: S-equol 10 mg BID vs S-equol 50 mg BID vs S-equol 150 mg BID vs Placebo; Severity of VMS per week at each protocol visits = (Sum of scores of Mild, Moderate, Severe hot flushes)/(Current protocol visit date-Previous protocol visit date (days)) x 7, where severity of vasomotor symptoms are scored as: 1 = mild, 2 = moderate and 3 = severe; Test type: Superiority or Other; p = 0.1609, Repeated measures ANCOVA — P-value was not adjusted for multiple comparisons and the a priori threshold for statistical significance was P <0.05. Treatment effect averaged across Weeks 1, 2 and 4; Mixed Model: Severity of VMS = Baseline (severity of VMS) + Treatment + Site + Weeks + Treatment x Weeks
Statistical Analysis 2: Comparison: S-equol 10 mg BID vs Placebo; Week 1, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = -6.34, 95% CI 2-sided [-26.41 to 13.73]
Statistical Analysis 3: Comparison: S-equol 50 mg BID vs Placebo; Week 1, Treatment Effect; Test type: Superiority or Other; p < 0.05, Pair-wise comparisons; LS means difference = 25.67, 95% CI 2-sided [5.64 to 45.69]
Statistical Analysis 4: Comparison: S-equol 150 mg BID vs Placebo; Week 1, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = 2.09, 95% CI 2-sided [-18.21 to 22.39]
Statistical Analysis 5: Comparison: S-equol 10 mg BID; Week 2, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = -16.14, 95% CI 2-sided [-43.29 to 11.01]
Statistical Analysis 6: Comparison: S-equol 50 mg BID vs Placebo; Week 2, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = 8.73, 95% CI 2-sided [-18.19 to 35.65]
Statistical Analysis 7: Comparison: S-equol 150 mg BID vs Placebo; Week 2, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = -0.65, 95% CI 2-sided [-27.80 to 26.50]
Statistical Analysis 8: Comparison: S-equol 10 mg BID vs Placebo; Week 4, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = -1.69, 95% CI 2-sided [-28.68 to 25.30]
Statistical Analysis 9: Comparison: S-equol 50 mg BID vs Placebo; Week 4, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = 16.15, 95% CI 2-sided [-10.40 to 42.71]
Statistical Analysis 10: Comparison: S-equol 150 mg BID vs Placebo; Week 4, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = -1.29, 95% CI 2-sided [-28.18 to 25.60]

5. Secondary Outcome: Change From Baseline (Day 0) in Vaginal pH at Week 2 and Week 4
Description: The pH scale measures how acidic or basic a substance is. The pH scale ranges from 0 to 14. A pH of 7 is neutral. A pH less than 7 is acidic. A pH greater than 7 is basic. The pH scale is logarithmic and as a result, each whole pH value below 7 is ten times more acidic than the next higher value.
  Normal vaginal pH is 3.8 to 4.5, slightly acidic.
  The LSMeans refer to overall adjusted mean pH.
Time Frame: 2 and 4 weeks from Baseline (Day 0)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo
Number analyzed (Participants) | 42 | 42 | 41 | 42
units on a scale
  Baseline (Day 0) | 5.5 [5.3 to 5.8] | 5.5 [5.3 to 5.8] | 5.8 [5.7 to 6.0] | 5.7 [5.5 to 6.0]
  Week 2 | 5.4 [5.2 to 5.6] | 5.4 [5.2 to 5.6] | 5.8 [5.5 to 6.1] | 5.8 [5.5 to 6.0]
  Change from Baseline at Week 2 | -0.1 [-0.3 to 0.1] | -0.1 [-0.3 to 0.1] | -0.0 [-0.3 to 0.3] | 0.0 [-0.2 to 0.3]
  Week 2, LSMean | 5.51 [5.28 to 5.75] | 5.49 [5.27 to 5.72] | 5.75 [5.53 to 5.98] | 5.72 [5.49 to 5.94]
  Week 4 | 5.4 [5.1 to 5.7] | 5.5 [5.3 to 5.8] | 5.6 [5.4 to 5.8] | 5.8 [5.5 to 6.1]
  Change from Baseline at Week 4 | -0.2 [-0.4 to 0.1] | -0.0 [-0.2 to 0.2] | -0.3 [-0.5 to -0.1] | 0.0 [-0.2 to 0.2]
  Week 4, LSMean | 5.48 [5.28 to 5.68] | 5.61 [5.42 to 5.80] | 5.50 [5.30 to 5.69] | 5.74 [5.55 to 5.93]
Statistical Analysis 1: Comparison: S-equol 10 mg BID vs S-equol 50 mg BID vs S-equol 150 mg BID vs Placebo; Test type: Superiority or Other; p = 0.2211, Repeated measures ANCOVA — P-value was not adjusted for multiple comparisons and the a priori threshold for statistical significance was P <0.05. Treatment effect averaged across Weeks 2 and 4; Mixed Model: (Vaginal pH) = Baseline (Vaginal pH) + Treatment + Site + Weeks + Treatment x Weeks
Statistical Analysis 2: Comparison: S-equol 10 mg BID vs Placebo; Week 2, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = -0.21, 95% CI 2-sided [-0.53 to 0.12]
Statistical Analysis 3: Comparison: S-equol 50 mg BID vs Placebo; Week 2, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = -0.23, 95% CI 2-sided [-0.55 to 0.09]
Statistical Analysis 4: Comparison: S-equol 150 mg BID vs Placebo; Week 2, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = 0.03, 95% CI 2-sided [-0.28 to 0.35]
Statistical Analysis 5: Comparison: S-equol 10 mg BID vs Placebo; Week 4, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = -0.26, 95% CI 2-sided [-0.54 to 0.02]
Statistical Analysis 6: Comparison: S-equol 50 mg BID vs Placebo; Week 4, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = -0.13, 95% CI 2-sided [-0.40 to 0.14]
Statistical Analysis 7: Comparison: S-equol 150 mg BID vs Placebo; Week 4, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = -0.24, 95% CI 2-sided [-0.51 to 0.03]

6. Secondary Outcome: Change From Baseline in Vaginal Maturation Index at Week 2 and Week 4
Description: The Vaginal Maturation Index was calculated by examining the maturation of the vaginal epithelium as adjudged by the cell types exfoliated. Parabasal cells are the least mature cells, intermediate cells display mild maturation, and superficial cells display the most maturity. The cell count is expressed as a percentage. The Vaginal Maturation Index was calculated as: 0.2*(parabasal cells, %)+0.6*(intermediate cells, %)+1.0*(superficial cells, %). This method is described in Menopause 2005;12(6):708-15.
  The index serves as an objective means of evaluating hormonal secretion or response; lower values indicate more immature cells on the surface (atrophy), while higher values indicate more mature epithelium.
  The LSMeans refer to overall adjusted mean percent of cells counted.
Time Frame: 2 and 4 weeks from Baseline (Day 0)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo
Number analyzed (Participants) | 42 | 42 | 41 | 42
percentage of cells
  Baseline (Day 0) | 52.6 [47.4 to 57.9] | 55.7 [50.7 to 60.7] | 50.9 [44.7 to 57.2] | 43.5 [37.4 to 49.6]
  Week 2 | 54.5 [49.0 to 60.1] | 54.3 [47.4 to 61.1] | 50.8 [43.1 to 58.6] | 47.0 [41.0 to 52.9]
  Change from Baseline at Week 2 | -0.7 [-3.8 to 2.4] | -1.3 [-8.4 to 5.9] | 0.6 [-6.5 to 7.7] | 3.9 [-3.0 to 10.8]
  Week 2, LSMean | 50.89 [45.29 to 56.50] | 50.89 [45.20 to 56.58] | 50.88 [45.09 to 56.67] | 52.47 [46.80 to 58.14]
  Week 4 | 56.5 [50.8 to 62.2] | 51.7 [45.5 to 57.9] | 51.3 [45.2 to 57.5] | 48.1 [42.2 to 54.0]
  Change from Baseline at Week 4 | 1.7 [-2.1 to 5.5] | -3.7 [-7.0 to -0.3] | 0.3 [-4.6 to 5.2] | 5.2 [-0.8 to 11.3]
  Week 4, LSMean | 53.58 [48.92 to 58.24] | 47.75 [43.35 to 52.14] | 51.01 [46.62 to 55.40] | 53.26 [49.52 to 58.26]
Statistical Analysis 1: Comparison: S-equol 10 mg BID vs S-equol 50 mg BID vs S-equol 150 mg BID vs Placebo; Vaginal maturation index = 0.2 x (% parabasal cells) + 0.6 x(% intermediate cells) + 1.0 x (% superficial cells); Test type: Superiority or Other; p = 0.6375, Repeated measures ANCOVA — [p-value comment as in outcome 5, analysis 1]; Mixed Model: (Vaginal Maturation Index) = Baseline (Vaginal Maturation Index) + Treatment + Site + Weeks + Treatment x Weeks
Statistical Analysis 2: Comparison: S-equol 10 mg BID vs Placebo; Week 2, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = -1.58, 95% CI 2-sided [-9.57 to 6.42]
Statistical Analysis 3: Comparison: S-equol 50 mg BID vs Placebo; Week 2, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = -1.58, 95% CI 2-sided [-9.63 to 6.46]
Statistical Analysis 4: Comparison: S-equol 150 mg BID; Week 2, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = -1.59, 95% CI 2-sided [-9.66 to 6.47]
Statistical Analysis 5: Comparison: S-equol 10 mg BID vs Placebo; Week 4, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = -0.31, 95% CI 2-sided [-6.73 to 6.11]
Statistical Analysis 6: Comparison: S-equol 50 mg BID vs Placebo; Week 4, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = -6.14, 95% CI 2-sided [-12.36 to 0.07]
Statistical Analysis 7: Comparison: S-equol 150 mg BID vs Placebo; Week 4, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = -2.88, 95% CI 2-sided [-9.05 to 3.28]

7. Secondary Outcome: Change From Baseline in Estradiol Concentration at Weeks 2 and 4
Description: The LSMeans refer to overall adjusted mean estradiol concentration.
Time Frame: 2 and 4 weeks from Baseline (Day 0)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Estradiol Concentration (pmol/L)
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo
Number analyzed (Participants) | 42 | 42 | 41 | 42
Estradiol Concentration (pmol/L)
  Baseline (Day 0) | 79.0 [55.5 to 102.5] | 65.7 [53.8 to 77.6] | 66.1 [53.1 to 79.2] | 59.6 [50.2 to 69.1]
  Week 2 | 117.3 [69.4 to 165.2] | 72.2 [54.4 to 90.1] | 68.1 [51.0 to 85.2] | 62.1 [51.1 to 73.1]
  Change from Baseline at Week 2 | 40.2 [-2.4 to 82.9] | 6.7 [-10.3 to 23.7] | 2.0 [-9.0 to 12.9] | 2.5 [-4.5 to 9.5]
  Week 2, LSMean | 104.93 [81.11 to 128.76] | 73.22 [49.98 to 96.46] | 65.03 [41.80 to 88.26] | 69.61 [46.24 to 92.99]
  Week 4 | 114.0 [48.1 to 179.9] | 82.8 [45.5 to 120.1] | 60.0 [45.2 to 74.7] | 70.4 [40.0 to 100.8]
  Change from Baseline at Week 4 | 37.5 [-8.4 to 83.4] | 20.3 [-18.5 to 59.2] | -6.7 [-19.1 to 5.6] | 10.7 [-18.3 to 39.8]
  Week 4, LSMean | 100.89 [67.96 to 133.81] | 86.56 [54.78 to 118.34] | 56.03 [24.14 to 87.91] | 78.77 [47.31 to 110.23]
Statistical Analysis 1: Comparison: S-equol 10 mg BID vs S-equol 50 mg BID vs S-equol 150 mg BID vs Placebo; Test type: Superiority or Other; p = 0.0681, Repeated measures ANCOVA — P-value is adjusted for multiple comparisons and the a priori threshold for statistical significance was P <0.05. Treatment effect averaged across Weeks 2 and 4; Mixed Model: (Estradiol) = Baseline (Estradiol) + Treatment + Site + Weeks + Treatment x Weeks
Statistical Analysis 2: Comparison: S-equol 10 mg BID vs Placebo; Week 2, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = 35.32, 95% CI 2-sided [1.75 to 68.90]
Statistical Analysis 3: Comparison: S-equol 50 mg BID vs Placebo; Week 2, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = 3.61, 95% CI 2-sided [-29.12 to 36.34]
Statistical Analysis 4: Comparison: S-equol 150 mg BID vs Placebo; Week 2, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = -4.58, 95% CI 2-sided [-37.39 to 28.23]
Statistical Analysis 5: Comparison: S-equol 10 mg BID vs Placebo; Week 4, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = 22.12, 95% CI 2-sided [-23.56 to 67.80]
Statistical Analysis 6: Comparison: S-equol 50 mg BID vs Placebo; Week 4, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = 7.80, 95% CI 2-sided [-36.70 to 52.29]
Statistical Analysis 7: Comparison: S-equol 150 mg BID vs Placebo; Week 4, Treatment Effect; Test type: Superiority or Other; p > 0.05, Pair-wise comparisons; LS means difference = -22.74, 95% CI 2-sided [-67.44 to 21.96]

8. Secondary Outcome: Change From Baseline in Progesterone Concentration at Week 2 and Week 4
Description: No repeated measures ANCOVA results are presented for change from Baseline in progesterone concentrations since the model did not converge.
Time Frame: 2 and 4 weeks from Baseline (Day 0)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Progesterone Concentration (nmol/L)
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo
Number analyzed (Participants) | 42 | 42 | 41 | 42
Progesterone Concentration (nmol/L)
  Baseline (Day 0) | 1.1 [1.0 to 1.3] | 1.1 [0.9 to 1.3] | 1.3 [0.9 to 1.6] | 1.1 [0.9 to 1.3]
  Week 2 | 1.2 [1.0 to 1.3] | 1.3 [1.0 to 1.5] | 1.1 [0.9 to 1.2] | 1.0 [0.9 to 1.2]
  Change from Baseline at Week 2 | 0.0 [-0.1 to 0.1] | 0.1 [-0.0 to 0.3] | -0.2 [-0.6 to 0.1] | -0.0 [-0.1 to 0.0]
  Week 4 | 7.0 [-4.8 to 18.9] | 1.1 [0.9 to 1.2] | 1.4 [0.8 to 2.0] | 1.1 [0.9 to 1.2]
  Change from Baseline at Week 4 | 5.9 [-5.9 to 17.8] | -0.0 [-0.1 to 0.0] | 0.1 [-0.2 to 0.4] | -0.0 [-0.1 to 0.0]

9. Secondary Outcome: Mean Change in the Menopause Rating Scale Total Score From Baseline at Week 4
Description: MRS consists of 11 menopause symptoms. The scoring scheme is simple, i.e., the score increases point by point with increasing severity of subjectively perceived symptoms in each of the 11 items (severity 0 [no complaints] 4 scoring points [extremely severe symptoms]). The respondent provides her personal perception by checking one of 5 possible boxes of "severity" for each of the items. The composite score (total score) is the sum of the 11 item scores, which can range from 0 (no symptoms) to 44 (extremely severe symptoms). Low total scores represent less severe menopause symptoms while higher scores represent more severe symptoms.
Time Frame: 4 weeks from Baseline (Day 0)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo
Number analyzed (Participants) | 42 | 42 | 41 | 42
units on a scale
  Baseline (Day 0) | 16.9 [14.3 to 19.5] | 17.3 [14.6 to 20.1] | 15.7 [13.3 to 18.1] | 14.5 [12.6 to 16.4]
  Week 4 | 11.5 [8.7 to 14.2] | 10.8 [8.5 to 13.1] | 9.7 [7.7 to 11.7] | 9.9 [8.3 to 11.6]
  Change from Baseline at Week 4 | -5.3 [-7.0 to 3.7] | -6.4 [-8.3 to 4.4] | -6.0 [-8.5 to 3.6] | -4.6 [-6.4 to 2.8]

10. Post Hoc Outcome: Change From Baseline in Menopause Rating Scale (MRS) - Sum of 3 Symptoms (Irritability, Dry Vagina, Joint/Muscular Discomfort)
Description: Note: Each MRS symptoms is assigned a score from 0 to 4 (0 = 'None' and 4 = 'Extremely severe').
  Scores for Symptoms 5, 10, and 11 on the MRS were summed and analyzed. Total summed scores ranged from 0 to 12, with higher scores representing more severe symptoms.
Time Frame: 4 weeks from Baseline (Day 0)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo
Number analyzed (Participants) | 42 | 42 | 41 | 42
units on a scale
  Baseline (Day 0) | 4.0 [3.2 to 4.9] | 4.2 [3.3 to 5.2] | 4.0 [3.2 to 4.8] | 3.4 [2.8 to 4.0]
  Week 4 | 2.8 [2.0 to 3.7] | 2.8 [2.1 to 3.6] | 2.5 [1.9 to 3.2] | 2.9 [2.3 to 3.5]
  Change from Baseline at Week 4 | -1.3 [-1.9 to -0.7] | -1.5 [-2.3 to -0.8] | -1.5 [-2.2 to -0.7] | -0.5 [-1.1 to 0.1]

11. Post Hoc Outcome: Percentage Change From Baseline in Menopause Rating Scale (MRS) - Sum of 3 Symptoms (Irritability, Dry Vagina, Joint/Muscular Discomfort)
Description: Percentage change from Baseline at Week 4 = (Week 4 value - Day 0 value)/(Day 0 value) x 100. Note: Each MRS symptoms is assigned a score from 0 to 4 (0 = 'None' and 4 = 'Extremely severe').
Time Frame: 4 weeks from Baseline (Day 0)
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo
Number analyzed (Participants) | 42 | 42 | 41 | 42
Percentage Change | -29.1 [-49.5 to -8.7] | -32.7 [-50.6 to -14.8] | -30.2 [-49.6 to -10.9] | -0.6 [-23.2 to 21.9]
Statistical Analysis 1: Comparison: S-equol 10 mg BID vs Placebo; Test type: Superiority or Other; p = 0.0475, Wilcoxon (Mann-Whitney) — P-value was not adjusted for multiple comparisons and the a priori threshold for statistical significance was P <0.05; Wilcoxon Mann-Whitney test: S-equol treatment group versus Placebo: Percentage Change from Baseline at Week 4
Statistical Analysis 2: Comparison: S-equol 50 mg BID vs Placebo; Test type: Superiority or Other; p = 0.0258, Wilcoxon (Mann-Whitney) — P-value was not adjusted for multiple comparisons and the a priori threshold for statistical significance P <0.05; Wilcoxon Mann-Whitney test: S-equol treatment group versus Placebo: Percentage Change from Baseline at Week 4
Statistical Analysis 3: Comparison: S-equol 150 mg BID vs Placebo; Test type: Superiority or Other; p = 0.0281, Wilcoxon (Mann-Whitney) — P-value was not adjusted for multiple comparisons and the a priori threshold for statistical significance was P <0.05; Wilcoxon Mann-Whitney test: S-equol treatment group versus Placebo: Percentage Change from Baseline at Week 4
Statistical Analysis 4: Comparison: S-equol 10 mg BID vs S-equol 50 mg BID vs S-equol 150 mg BID vs Placebo; All three S-equol treatment arms were aggregated and compared to placebo; Test type: Superiority or Other; p = 0.0645, Kruskal-Wallis

12. Post Hoc Outcome: Change From Baseline in Menopause Rating Scale (MRS) - Sum of 3 Symptoms (Irritability, Dry Vagina, Joint/Muscular Discomfort) - S-equol Groups Combined
Description: The following analysis shows the results when the S-equol groups (S-equol 20 mg total daily dose, 100 mg total daily dose, and 300 mg total daily dose) are combined and regarded as a single treatment group.
  Note: Each MRS symptoms was assigned a score from 0 to 4 (0 = 'None' and 4 = 'Extremely severe'
Time Frame: 4 weeks from Baseline (Day 0)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- S-equol Groups Combined: The S-equol groups (S-equol 20 mg total daily dose, 100 mg total daily dose, and 300 mg total daily dose) were combined and regarded as a single treatment group.
Arm/Group | S-equol Groups Combined | Placebo
Number analyzed (Participants) | 125 | 42
units on a scale
  Baseline (Day 0) | 4.1 [3.6 to 4.6] | 3.4 [2.8 to 4.0]
  Week 4 | 2.7 [2.3 to 3.2] | 2.9 [2.3 to 3.5]
  Change from Baseline at Week 4 | -1.4 [-1.8 to -1.0] | 0.0 [-1.1 to 0.1]
Statistical Analysis 1: Comparison: S-equol Groups Combined vs Placebo; Test type: Superiority or Other; p = 0.0097, Wilcoxon (Mann-Whitney) — P-value is adjusted for multiple comparisons and the a priori threshold for statistical significance was P <0.05; Wilcoxon Mann-Whitney test: S-equol groups combined versus Placebo: Change from Baseline at Week 4

13. Secondary Outcome: Mean Precentage Change in the Menopause Rating Scale Total Score From Baseline at Week 4
Description: Percentage change from Baseline at Week 4 = (Week 4 value - Day 0 value)/(Day 0 value) x 100. Note: MRS consists of 11 symptoms, where each symptom is assigned a score from 0 to 4 (0 = 'None' and 4 = 'Extremely severe').
Time Frame: 4 weeks from Baseline (Day 0)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo
Number analyzed (Participants) | 42 | 42 | 41 | 42
Percentage Change | -36.7 [-46.8 to -26.6] | -37.4 [-46.9 to -27.9] | -30.6 [-43.8 to -17.4] | -27.4 [-39.2 to 15.6]
Statistical Analysis 1: Comparison: S-equol 10 mg BID vs Placebo; Test type: Superiority or Other; p = 0.4352, Wilcoxon (Mann-Whitney) — P-value was not adjusted for multiple comparisons and the a priori threshold for statistical significance was P <0.05; Wilcoxon Mann-Whitney test: S-equol treatment group versus Placebo: Percentage Change from Baseline at Week 4
Statistical Analysis 2: Comparison: S-equol 50 mg BID vs Placebo; Test type: Superiority or Other; p = 0.2600, Wilcoxon (Mann-Whitney) — P-value was not adjusted for multiple comparisons and the a priori threshold for statistical significance was P <0.05; Wilcoxon Mann-Whitney test: S-equol treatment group versus Placebo: Percentage Change from Baseline at Week 4
Statistical Analysis 3: Comparison: S-equol 150 mg BID vs Placebo; Test type: Superiority or Other; p = 0.7037, Wilcoxon (Mann-Whitney) — P-value was not adjusted for multiple comparisons and the a priori threshold for statistical significance was P <0.05; Wilcoxon Mann-Whitney test: S-equol treatment group versus Placebo: Percentage Change from Baseline at Week 4
Statistical Analysis 4: Comparison: S-equol 10 mg BID vs S-equol 50 mg BID vs S-equol 150 mg BID vs Placebo; All three S-equol treatment arms were aggregated and compared to placebo; Test type: Superiority or Other; p = 0.7155, Kruskal-Wallis

14. Post Hoc Outcome: Change From Baseline in Menopause Rating Scale (MRS) - Dryness of Vagina- S-equol Groups Combined
Description: The following analysis pre-specified the combining of all S-equol groups (S-equol 20 mg total daily dose, 100 mg total daily dose, and 300 mg total daily dose) into a single treatment group. The results from the Wilcoxon-Mann-Whitney test (pair-wise test), based on the change from Baseline at Week 4, are presented.
  Note: Dryness of Vagina was assigned a score from 0 to 4 (0 = 'None' and 4 = 'Extremely severe'
Time Frame: 4 weeks from Baseline (Day 0)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | S-equol Groups Combined | Placebo
Number analyzed (Participants) | 125 | 42
units on a scale
  Baseline (Day 0) | 1.5 [1.2 to 1.7] | 1.5 [1.1 to 1.9]
  Week 4 | 1.1 [0.8 to 1.3] | 1.4 [1.0 to 1.8]
  Change from Baseline at Week 4 | -0.4 [-0.6 to -0.3] | -0.1 [-0.4 to 0.2]
Statistical Analysis 1: Comparison: S-equol Groups Combined vs Placebo; Test type: Superiority or Other; p = 0.0381, Wilcoxon (Mann-Whitney) — P-value is adjusted for multiple comparisons and the a priori threshold for statistical significance was P <0.05; Wilcoxon Mann-Whitney test: S-equol groups combined versus Placebo: Change from Baseline at Week 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of signing of the informed consent document through the follow-up visit or early termination visit (whichever occurred first).
Description: An adverse event was followed to a satisfactory resolution, until it became stable, or until it could be explained by another known cause(s) and clinical judgment indicated that further evaluation was not warranted, or 30 days from the date of last study drug dose for adverse events not related to study drug.
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo
Serious Adverse Events (participants affected / at risk) | 1/43 | 0/42 | 1/42 | 0/42
Other Adverse Events (participants affected / at risk) | 20/43 | 20/42 | 17/42 | 15/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S-equol 10 mg BID (N=43) | S-equol 50 mg BID (N=42) | S-equol 150 mg BID (N=42) | Placebo (N=42)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S-equol 10 mg BID (N=43) | S-equol 50 mg BID (N=42) | S-equol 150 mg BID (N=42) | Placebo (N=42)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac Disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Abnormal Feces (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (7) | 3 (3) | 3 (3) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection Site Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irritability (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune System Disorders (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal Allergy (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oral Herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 2 (2) | 6 (6) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 2 (2) | 3 (3) | 0 (0)
Vaginal Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint Sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Mouth Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural Hypertension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Glucose Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Lactate Dehydrogenase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Triglycerides Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Estradiol Increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Smear Cervix Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Migraine (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mood Swings (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast Tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical Dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometrial Hypertrophy (Reproductive system and breast disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Vaginal Discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Vulvovaginal Erythema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash Macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Hypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot Flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Per-protocol, an ANOVA model was to be used for the primary efficacy analysis. However using statistical adjustment of baseline values, ANCOVA could be more a more powerful analysis (Vickers AJ. BMC Med Res Methodology. 2001;1:6. Epub 2001 Jun 28).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less